CLINICAL TRIAL: NCT05724316
Title: Open Controlled Trial to Explore the Effectiveness of Vitamin D Supplements on the Behaviours, Mental, and Physical Health of United Kingdom Prison Residents
Brief Title: Effects of Vitamin D on the Behaviours, Mental, and Physical Health of Prisoners
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oxford Brookes University (Other)
Collaborators: HM Prison and Probation Service, United Kingdom (Unknown); Ministry of Justice, United Kingdom (Unknown); University of Oxford (Other); Practice Plus Group (Unknown)
Responsible Party: Principal Investigator, Jonathan Tammam, Director Centre for Nutrition and Health, Oxford Brookes University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 221634
Record Dates: First submitted 2022-12-21; First posted 2023-02-13 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-11

CONDITIONS: Mental Wellbeing; Depression, Anxiety; Bone Density, Low; Vitamin D Deficiency; Behavior
Keywords: Anxiety; Depression; Behaviour; Mental health; Mental wellbeing; Physical health; Bone health; Prisoners
MeSH Terms: conditions — Depression; Anxiety Disorders; Bone Diseases, Metabolic; Vitamin D Deficiency; Behavior; Psychological Well-Being | interventions — Cholecalciferol; Tablets

STUDY DESIGN:
Intervention Model Description: One arm will receive vitamin D supplements, the other arm will not receive supplements.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D Group (Experimental): All participants in this group will receive cholecalciferol (VD3 25μg) tablets, one to be taken per day.
  Interventions: Dietary Supplement: Vitamin D supplement
- Control Group (No Intervention): Will receive no vitamin D supplements.

INTERVENTIONS:
Dietary Supplement: Vitamin D supplement — N/A (says not to repeat information here)
  Other Names: cholecalciferol (VD3 25μg) tablet
  Arms: Vitamin D Group

SUMMARY:
This study aims to understand how vitamin D (VD) affects human health. Typically, prisoners are low on vitamin D, as it is difficult to receive through diet, and is mostly obtained via exposure to the sun. The investigators predict that VD supplements could help improve overall mental well-being, as well as improve bone health. The investigators aim to recruit two groups of participants from a United Kingdom (UK) Prison, all of whom will participate via an informed consent process. The first group of prisoners will have chosen to take VD supplements, the second group will have chosen not to take VD supplements. At the start of the study, prisoners will have their bone density and blood VD levels tested. The investigators will also ask participants to complete a series of questionnaires to understand the state of mental well-being at the start of the study. Participants will be asked to complete a food diary to track dietary intake over the following week. Additionally, the investigators are interested in identifying what proportion of participants have a specific genetic makeup relating to their ability to metabolise VD, and participants will be asked to provide a saliva sample to test this. Every month following the start of the study, participants will be asked to complete the same questionnaires and food diary again. On the 3rd month, the investigators will again test the participants' bone density and blood levels of VD, to see whether supplementation has improved participant VD status. This study will run for a minimum of 3 months, up to a maximum of 6.

DETAILED DESCRIPTION:
Aim of this research:

This is a quantitative open-label controlled trial, aiming to assess the effect of VD supplementation, within offender populations (male adults 21+), on behaviours, physical and mental health outcomes.

Primary Aims:

1. To assess the prevalence of VD supplementation within prisons.
2. To assess VD serum levels among male adult prisoner population.
3. To assess whether VD supplementation in prisons can lead to improved markers of physical health, for example, grip strength, bone density.
4. To assess whether VD supplementation in prisons can lead to an overall improvement of mental health wellbeing, including anxiety and depression severity, assessed using validated methods.
5. To assess whether VD can lead to improved behaviour amongst prisoners, assessed using a self-reported aggression questionnaire, and governor adjudication reports.

Secondary Aims:

1. To determine whether aim 2 is associated with individual differences in VD metabolism.
2. To assess overall nutritional content and quality of prison dietary intake.

This research has five hypotheses:

1. VD supplementation will improve Serum 25-hydroxyvitamin D (VD) levels.
2. VD supplementation will reduce levels of anxiety and depression within the offender population (measured by GAD-7 and PHQ-9).
3. VD will improve general mental well-being (measured by WEMWBS).
4. VD supplementation will improve physical health outcomes within the offender population (measured by VD blood serum level, bone density, and grip strength)
5. VD supplementation will reduce violence and aggressive behaviours (measured by Buss Perry AQ, and adjudication reports)

Study Design:

A minimum of 100 participants (50 per group) will be sought for recruitment (+10% for attrition). The sample size is based on The Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS) which ideally recommends a minimum of 50 participants per group (100 total) to detect a difference of +/- 5 points. This sample size is calculated using a power of 0.8, at a significance level of 0.05.

Group 1 (experimental group) will be supplemented with VD (1x25ug VD3 cholecalciferol tablet per day), and group 2 will not be supplemented with VD (control group). Upon recruitment, participants will be identified as either taking VD, or not. Participants taking VD will be in Group 1, participants not taking VD will be in Group2 (control).

Baseline Measures:

From Participant:

1. Demographic information: (age, sex, ethnicity/race, gender, level of education, custodial status and length)
2. Health measures: (height, weight, body mass index (BMI), grip strength)
3. Dietary intake: food diary (7-day food diary will be provided to participants)
4. Self-Reported Questionnaires: Patient Health Questionnaire-9 (PHQ-9) (for depression), Generalised Anxiety Disorder Assessment (GAD-7) (for anxiety), Buss Perry Aggression Questionnaire (AQ) (for aggression), and WEMWBS (for general mental wellbeing)
5. A survey question regarding time spent outside on average, and the date participant first took supplement (if applicable)
6. Bone density
7. Blood analysis (for VD serum) (researcher will be qualified for blood-taking procedures)
8. Saliva analysis (for genetics)

From Prison

1. Health history (including medications taking)
2. Behaviour records (governor/officer reports, adjudication reports)
3. Mental health history (i.e. any diagnoses/treatment for depression, anxiety, bipolar, schizophrenia, any reports of self-harm/suicide attempts)
4. Substance use (any misuse history)
5. Dietary issues (history of hunger strikes)
6. Date of resident entry to prison and length of stay

After baseline, the following measures will be taken at the end of month 1 and month 2:

From Participant:

1. Questionnaires: PHQ-9, GAD-7, AQ, and WEMWBS
2. Log/Question regarding time spent outside

At the end of month 3, the following measures will be taken:

From Participant:

1. Blood analysis: Serum 25-hydroxyvitamin D (25(OH)D)
2. Bone density
3. Grip strength
4. Weight, height, and BMI
5. 3- or 7-day food diary (will depend on what is discussed with identified prisons)

And the regular monthly measures:

1. Questionnaires: PHQ-9, GAD-7, AQ, and WEMWBS
2. Log/Question regarding time spent outside

ELIGIBILITY:
Inclusion Criteria:

* Long-term Residents (with minimum 1 year)
* Biological Male adults (+18)
* Have been residents for minimum of 3 months
* Understanding of the English language

Exclusion Criteria:

* Short term Residents (<1 year), residents at end of their sentence
* Residents with conditions impacting nutrient absorption i.e. Crohn's disease/celiac disease
* Residents already taking calcitriol (an active form of VD)
* Any medical condition that would preclude a participant from taking VD supplements
* Any medical condition which could interfere with VD metabolism

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2023-03-18 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Mental wellbeing | Baseline
  Overall mental well-being as measured by The Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS).
  WEMWBS uses a five-point scale, with participants required to answer questions recalling from the previous 2 weeks. The minimum score is 14, the maximum score is 70. A high score indicates lower well-being.
Mental wellbeing | End of Month 1
  Overall mental well-being as measured by The Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS).
  WEMWBS uses a five-point scale, with participants required to answer questions recalling from the previous 2 weeks. The minimum score is 14, the maximum score is 70. A high score indicates lower well-being.
Mental wellbeing | End of Month 2
  Overall mental well-being as measured by The Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS).
  WEMWBS uses a five-point scale, with participants required to answer questions recalling from the previous 2 weeks. The minimum score is 14, the maximum score is 70. A high score indicates lower well-being.
Mental wellbeing | End of Month 3
  Overall mental well-being as measured by The Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS).
  WEMWBS uses a five-point scale, with participants required to answer questions recalling from the previous 2 weeks. The minimum score is 14, the maximum score is 70. A high score indicates lower well-being.
Vitamin D serum levels | Baseline
  Assessing the levels of serum vitamin D amongst participants, using blood serum. 25(OH)D of < 20 ng/ml is considered vitamin D deficiency, and 25(OH)D of 21-29 ng/ml is considered insufficient.
Vitamin D serum levels | End of month 3
  Assessing the levels of serum vitamin D amongst participants, using blood serum. 25(OH)D of < 20 ng/ml is considered vitamin D deficiency, and 25(OH)D of 21-29 ng/ml is considered insufficient.

SECONDARY OUTCOMES:
Rule Violations | Baseline
  Measured by officer/governor reports and adjudication reports.
Rule Violations | End of Month 3
  Measured by officer/governor reports and adjudication reports.
Aggression | Baseline
  Aggression is measured by Buss-Perry Aggression Questionnaire (AQ). The Buss-Perry AQ consists of 34 statements, which participants answer recalling from the previous 2 weeks. Higher T-scores indicate a higher level of aggression. Participants rate each statement using a 5-point Likert scale. Scores are normalised to a scale of 0-1, with 1 representing the highest level of aggression.
Aggression | End of Month 1
  Aggression is measured by Buss-Perry Aggression Questionnaire (AQ). The Buss-Perry AQ consists of 34 statements, which participants answer recalling from the previous 2 weeks. Higher T-scores indicate a higher level of aggression. Participants rate each statement using a 5-point Likert scale. Scores are normalised to a scale of 0-1, with 1 representing the highest level of aggression.
Aggression | End of Month 2
  Aggression is measured by Buss-Perry Aggression Questionnaire (AQ). The Buss-Perry AQ consists of 34 statements, which participants answer recalling from the previous 2 weeks. Higher T-scores indicate a higher level of aggression. Participants rate each statement using a 5-point Likert scale. Scores are normalised to a scale of 0-1, with 1 representing the highest level of aggression.
Aggression | End of Month 3
  Aggression is measured by Buss-Perry Aggression Questionnaire (AQ). The Buss-Perry AQ consists of 34 statements, which participants answer recalling from the previous 2 weeks. Higher T-scores indicate a higher level of aggression. Participants rate each statement using a 5-point Likert scale. Scores are normalised to a scale of 0-1, with 1 representing the highest level of aggression.
Generalised anxiety | Baseline
  Generalised anxiety disorder as measured by GAD-7. The minimum score is 0, the highest is 21. A higher score indicates higher levels of generalised anxiety.
Generalised anxiety | End of Month 1
  Generalised anxiety disorder as measured by GAD-7. The minimum score is 0, the highest is 21. A higher score indicates higher levels of generalised anxiety.
Generalised anxiety | End of Month 2
  Generalised anxiety disorder as measured by GAD-7. The minimum score is 0, the highest is 21. A higher score indicates higher levels of generalised anxiety.
Generalised anxiety | End of Month 3
  Generalised anxiety disorder as measured by GAD-7. The minimum score is 0, the highest is 21. A higher score indicates higher levels of generalised anxiety.
Depression severity | Baseline
  Depression severity as measured by PHQ-9. Minimum score is 0, with the maximum of 27. A higher score indicates higher levels of depression.
Depression severity | End of Month 1
  Depression severity as measured by PHQ-9. Minimum score is 0, with the maximum of 27. A higher score indicates higher levels of depression.
Depression severity | End of Month 2
  Depression severity as measured by PHQ-9. Minimum score is 0, with the maximum of 27. A higher score indicates higher levels of depression.
Depression severity | End of Month 3
  Depression severity as measured by PHQ-9. Minimum score is 0, with the maximum of 27. A higher score indicates higher levels of depression.
Bone density | Baseline
  Bone density measured by Sonost 3000 bone densimeter.
Bone density | End of Month 3
  Bone density measured by Sonost 3000 bone densimeter.
Grip Strength | Baseline
  Grip strength as measured by a Takei Hand Grip Dynamometer.
Grip Strength | End of Month 3
  Grip strength as measured by a Takei Hand Grip Dynamometer.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Tammam, Principal Investigator — Oxford Brookes University
Locations (1):
- HMP Huntercombe, Henley on Thames, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Due to the nature of the participants included, we are undecided on whether raw data will be shared at this time. This will be reviewed later on with the collaborators.